CLINICAL TRIAL: NCT04617119
Title: The Effects of Multi-modality Physiotherapy in Delaying or Preventing COVID-19 Patient From Admitting to ICU: A Pilot Study
Brief Title: The Effects of Multi-modality Physiotherapy in Delaying or Preventing COVID-19 Patient From Admitting to ICU
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: DR. JASSIM ALGHAITH (Other Government)
Responsible Party: Sponsor-Investigator, DR. JASSIM ALGHAITH, Specialist physical therapist, PhD., Ministry of Health, Kuwait
Organization: Ministry of Health, Kuwait (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JALGHAITH
Record Dates: First submitted 2020-10-28; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Severe Systemic Illness Respiratory Muscle Fatigue
Keywords: Respiratory muscle strength; Inspiratory muscle training; Respiratory physical therapy; Patient exercise training; Maximal inspiratory pressure
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A pilot study following a randomized controlled trial design.
Who Masked: Participant, Outcomes Assessor
Masking Description: COVID-19 patient will be blinded from the study aim. The outcomes assessor will be blinded from the study aim and patient allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional physical therapy treatment and IMT (Experimental): The conventional physical therapy treatment for COVID-19 patient will be based on patient medical and physical status.
  In addition, the patient will receive inspiratory muscle training (IMT) by using a threshold IMT device. Patient will ask to use the device twice daily. In each time, patient will perform 3 sets of 10 breaths with 1-minute rest between sets.
  Exercise intensity will start with 10 % of pre-measured maximal inspiratory pressure.
  Once the patient successfully completed 30 breath twice a day, the exercise load will increase 5% more in the subsequent training session.
  This treatment protocol will perform daily for 2 weeks.
  Interventions: Device: Threshold IMT device; Other: Conventional physical therapy
- Conventional physical therapy (Active Comparator): The conventional physical therapy treatment for COVID-19 patient will be based on patient medical and physical status.
  Interventions: Other: Conventional physical therapy

INTERVENTIONS:
Device: Threshold IMT device — 10 breaths X 3 sets, two times a day for 2 weeks. starting intensity 10 % of pre-measured maximal inspiratory pressure.
  Arms: Conventional physical therapy treatment and IMT
Other: Conventional physical therapy — daily

SUMMARY:
This study aims to evaluate the effectiveness of respiratory muscle training with COVID-19 patient, who has underlying health conditions, in order to delay or prevent them from admitting to ICU.

ELIGIBILITY:
Inclusion Criteria:

* Non- intubated patient diagnosed with moderate to severe pneumonia (confirmed by chest x-ray and officially reported) as secondary to COVID-19 with one more symptom such as:

  1. Respiratory rate at ≥ 20 breath.min-1.
  2. Oxygen saturation (SatO2) ≤ 90% at rest on room air.
  3. Arterial partial pressure of oxygen (PaO2) ≤ 80 mmHg at resting.
  4. PaO2/FiO2 ratio or P/F (is the ratio between the arterial partial pressure of oxygen and the percentage of oxygen supplied) < 300mmHg.

Exclusion Criteria:

1. Patient that has received upper abdominal or thoracic surgery recently (≤ 3 months).
2. Cancer patients.
3. Pregnant patients.
4. Patient mentally unstable.
5. Patient with unstable cardiovascular or neurological functions.
6. Patients refusing to participate in this clinical trial.
7. Patient less the 21 years old (According to Kuwaiti Law).
8. Patients who have a language barrier who cannot understand Arabic or English.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2021-02-06 (Estimated); Study Completion 2021-04-06 (Estimated)

PRIMARY OUTCOMES:
Changes in Respiratory muscle performance | Baseline, 1st week, 2nd week, one month
  Changes in Respiratory muscle performance will be determined by using the Respiratory Pressure Meter device. Patient will perform full inspiration through this device for 1.5 seconds via the mouth (nose occluded). The reading of the negative peak pressure that is maintained for 1 second in the device is a maximal inspiration peak.

SECONDARY OUTCOMES:
Blood pressure | Daily from baseline to hospital discharge (2 weeks)
  Blood pressure measured by electronic BP machine before and after session
Heart rate | Daily from baseline to hospital discharge (2 weeks)
  measured by heart rate monitor before and after session
Oxygen saturation | Daily from baseline to hospital discharge (2 weeks)
  Measured by pulse oximeter before and after session
Oxygen supplementation | Daily from baseline to hospital discharge (2 weeks).
  Number of % of oxygen patient on it before and after session
Oxygen flow rate | Daily from baseline to hospital discharge (2 weeks)
  measuring the number of time where the oxygen above or below 4L/min.
Dyspnoea level | Daily from baseline to hospital discharge (2 weeks)
  By using Borg scale (rating of perceived exertion scale), Possible score range from 0 (nothing) to 10 ( Maximal exertion).
  Before and after session.
Pain level | Daily from baseline to hospital discharge (2 weeks)
  By using visual analogue scale. Possible score range from 0 (no pain) to 10 (worst possible pain) Before and after session.
Respiratory rate | Daily from baseline to hospital discharge (2 weeks)
  Measured by Respiratory rate monitor. Before and after session
Threshold IMT device | Daily from baseline to 1 month from admission
  Recording number for breath and sets daily.

CONTACTS AND LOCATIONS:
Locations (1):
- Jaber Al-Ahmed Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Background] WHO, CORONAVIRUS DISEASE (COVID-19) OUTBREAK: RIGHTS, ROLES AND RESPONSIBILITIES OF HEALTH WORKERS, INCLUDING KEY CONSIDERATIONS FOR OCCUPATIONAL SAFETY AND HEALTH 2020.
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Cascella M, Rajnik M, Aleem A, Dulebohn SC, Di Napoli R. Features, Evaluation, and Treatment of Coronavirus (COVID-19). 2023 Aug 18. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK554776/ PMID 32150360
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Arentz M, Yim E, Klaff L, Lokhandwala S, Riedo FX, Chong M, Lee M. Characteristics and Outcomes of 21 Critically Ill Patients With COVID-19 in Washington State. JAMA. 2020 Apr 28;323(16):1612-1614. doi: 10.1001/jama.2020.4326. PMID 32191259
- [Background] Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020 Apr 14;323(14):1335. doi: 10.1001/jama.2020.4344. No abstract available. PMID 32181795
- [Background] Zhou F, Yu T, Du R, Fan G, Liu Y, Liu Z, Xiang J, Wang Y, Song B, Gu X, Guan L, Wei Y, Li H, Wu X, Xu J, Tu S, Zhang Y, Chen H, Cao B. Clinical course and risk factors for mortality of adult inpatients with COVID-19 in Wuhan, China: a retrospective cohort study. Lancet. 2020 Mar 28;395(10229):1054-1062. doi: 10.1016/S0140-6736(20)30566-3. Epub 2020 Mar 11. PMID 32171076
- [Background] Honce R, Schultz-Cherry S. Impact of Obesity on Influenza A Virus Pathogenesis, Immune Response, and Evolution. Front Immunol. 2019 May 10;10:1071. doi: 10.3389/fimmu.2019.01071. eCollection 2019. PMID 31134099
- [Background] Bhatraju PK, Ghassemieh BJ, Nichols M, Kim R, Jerome KR, Nalla AK, Greninger AL, Pipavath S, Wurfel MM, Evans L, Kritek PA, West TE, Luks A, Gerbino A, Dale CR, Goldman JD, O'Mahony S, Mikacenic C. Covid-19 in Critically Ill Patients in the Seattle Region - Case Series. N Engl J Med. 2020 May 21;382(21):2012-2022. doi: 10.1056/NEJMoa2004500. Epub 2020 Mar 30. PMID 32227758
- [Background] Cai Q, Chen F, Wang T, Luo F, Liu X, Wu Q, He Q, Wang Z, Liu Y, Liu L, Chen J, Xu L. Obesity and COVID-19 Severity in a Designated Hospital in Shenzhen, China. Diabetes Care. 2020 Jul;43(7):1392-1398. doi: 10.2337/dc20-0576. Epub 2020 May 14. PMID 32409502
- [Background] Almazeedi S, Al-Youha S, Jamal MH, Al-Haddad M, Al-Muhaini A, Al-Ghimlas F, Al-Sabah S. Characteristics, risk factors and outcomes among the first consecutive 1096 patients diagnosed with COVID-19 in Kuwait. EClinicalMedicine. 2020 Jul 4;24:100448. doi: 10.1016/j.eclinm.2020.100448. eCollection 2020 Jul. PMID 32766546
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Laveneziana P, Albuquerque A, Aliverti A, Babb T, Barreiro E, Dres M, Dube BP, Fauroux B, Gea J, Guenette JA, Hudson AL, Kabitz HJ, Laghi F, Langer D, Luo YM, Neder JA, O'Donnell D, Polkey MI, Rabinovich RA, Rossi A, Series F, Similowski T, Spengler CM, Vogiatzis I, Verges S. ERS statement on respiratory muscle testing at rest and during exercise. Eur Respir J. 2019 Jun 13;53(6):1801214. doi: 10.1183/13993003.01214-2018. Print 2019 Jun. PMID 30956204
- [Background] Sood A. Altered resting and exercise respiratory physiology in obesity. Clin Chest Med. 2009 Sep;30(3):445-54, vii. doi: 10.1016/j.ccm.2009.05.003. PMID 19700043
- [Background] Castro AA, Calil SR, Freitas SA, Oliveira AB, Porto EF. Chest physiotherapy effectiveness to reduce hospitalization and mechanical ventilation length of stay, pulmonary infection rate and mortality in ICU patients. Respir Med. 2013 Jan;107(1):68-74. doi: 10.1016/j.rmed.2012.09.016. Epub 2012 Oct 22. PMID 23085215
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Dimitriadis Z, Kapreli E, Konstantinidou I, Oldham J, Strimpakos N. Test/retest reliability of maximum mouth pressure measurements with the MicroRPM in healthy volunteers. Respir Care. 2011 Jun;56(6):776-82. doi: 10.4187/respcare.00783. Epub 2011 Feb 9. PMID 21310113
- [Background] Ferraro FV, Gavin JP, Wainwright T, McConnell A. The effects of 8 weeks of inspiratory muscle training on the balance of healthy older adults: a randomized, double-blind, placebo-controlled study. Physiol Rep. 2019 May;7(9):e14076. doi: 10.14814/phy2.14076. PMID 31074198
- [Background] Alderson LM, Joksaite SX, Kemp J, Main E, Watson T, Platt FM, Cortina-Borja M. Age-related gait standards for healthy children and young people: the GOS-ICH paediatric gait centiles. Arch Dis Child. 2019 Aug;104(8):755-760. doi: 10.1136/archdischild-2018-316311. Epub 2019 Mar 25. PMID 30910816
- [Background] Jalan NS, Daftari SS, Retharekar SS, Rairikar SA, Shyam AM, Sancheti PK. Intra- and inter-rater reliability of maximum inspiratory pressure measured using a portable capsule-sensing pressure gauge device in healthy adults. Can J Respir Ther. 2015 Spring;51(2):39-42. PMID 26089737
- [Background] Remuzzi A, Remuzzi G. COVID-19 and Italy: what next? Lancet. 2020 Apr 11;395(10231):1225-1228. doi: 10.1016/S0140-6736(20)30627-9. Epub 2020 Mar 13. PMID 32178769
- [Background] Cai H. Sex difference and smoking predisposition in patients with COVID-19. Lancet Respir Med. 2020 Apr;8(4):e20. doi: 10.1016/S2213-2600(20)30117-X. Epub 2020 Mar 11. No abstract available. PMID 32171067
- [Background] Chiappa GR, Roseguini BT, Vieira PJ, Alves CN, Tavares A, Winkelmann ER, Ferlin EL, Stein R, Ribeiro JP. Inspiratory muscle training improves blood flow to resting and exercising limbs in patients with chronic heart failure. J Am Coll Cardiol. 2008 Apr 29;51(17):1663-71. doi: 10.1016/j.jacc.2007.12.045. PMID 18436118
- [Background] Edwards AM, Maguire GP, Graham D, Boland V, Richardson G. Four weeks of inspiratory muscle training improves self-paced walking performance in overweight and obese adults: a randomised controlled trial. J Obes. 2012;2012:918202. doi: 10.1155/2012/918202. Epub 2012 Jun 26. PMID 22792448
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Souza H, Rocha T, Pessoa M, Rattes C, Brandao D, Fregonezi G, Campos S, Aliverti A, Dornelas A. Effects of inspiratory muscle training in elderly women on respiratory muscle strength, diaphragm thickness and mobility. J Gerontol A Biol Sci Med Sci. 2014 Dec;69(12):1545-53. doi: 10.1093/gerona/glu182. PMID 25395284